CLINICAL TRIAL: NCT02790515
Title: Provision of TCRγδ T Cells and Memory T Cells Plus Selected Use of Blinatumomab in Naïve T-cell Depleted Haploidentical Donor Hematopoietic Cell Transplantation for Hematologic Malignancies Relapsed or Refractory Despite Prior Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REF2HCT; NCI-2016-00812 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myeloid Sarcoma; Chronic Myeloid Leukemia (CML); Juvenile Myelomonocytic Leukemia (JMML); Myelodysplastic Syndrome (MDS); Non-Hodgkin Lymphoma (NHL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Sarcoma, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; thymoglobulin; blinatumomab; Cyclophosphamide; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Filgrastim; Melphalan; Mesna; Rituximab; Tacrolimus; Thiotepa; Transplantation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Participants receive a conditioning regimen of antithymocyte globulin (rabbit), cyclophosphamide, mesna, fludarabine, thiotepa, tacrolimus (first 5 participants enrolled), sirolimus (used beginning with 6th enrolled participant), melphalan, rituximab. This is followed by HPC,A infusion (transplant), then by G-CSF and blinatumomab.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Anti-thymocyte globulin (rabbit); Drug: Blinatumomab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: G-CSF; Drug: Melphalan; Drug: Mesna; Drug: Rituximab; Drug: Tacrolimus; Drug: Thiotepa; Biological: HPC,A Infusion; Device: CliniMACS; Drug: Sirolimus

INTERVENTIONS:
Drug: Anti-thymocyte globulin (rabbit) — Given intravenous (IV) prior to transplant on Days -14, -13, -12.
  Other Names: Thymoglobulin®; rabbit ATG
Drug: Blinatumomab — Given by continuous IV infusion at least 2 weeks post-engraftment. Blinatumomab will be given only to patients with CD19+ malignancies.
  Other Names: Blincyto
Drug: Cyclophosphamide — Given by IV infusion prior to transplant on Day -9.
  Other Names: Cytoxan
Drug: Fludarabine — Given IV prior to transplant on Days -8, -7, -6, -5, and -4.
  Other Names: Fludara
Drug: G-CSF — Given IV or subcutaneous (SQ) following transplant on Days 6 and 7.
  Other Names: Filgrastim; Neupogen®
Drug: Melphalan — Given IV prior to transplant on Days -2 and -1.
  Other Names: L-phenylalanine mustard; Phenylalanine mustard; L-PAM; L-sarcolysin; Alkeran
Drug: Mesna — Given IV prior to cyclophosphamide administration and at approximately 3, 6, and 9 hours after cyclophosphamide infusion.
  Other Names: Mesnex
Drug: Rituximab — Given IV prior to transplant on Day -1.
  Other Names: Rituxan™
Drug: Tacrolimus — Given oral (PO) or IV beginning prior to transplant on Day -2. The dose will begin to taper at approximately day +60 after transplant in the absence of GVHD. Tacrolimus was used for the first 5 participants enrolled on study. Subsequent participants receive sirolimus.
  Other Names: FK506; Prograf®; Protopic®
Drug: Thiotepa — Given IV prior to transplant on Day -3.
  Other Names: Thioplex® by Immunex; TESPA; TSPA
Biological: HPC,A Infusion — Hematopoietic Progenitor Cell, Apheresis (HPC,A) infusion of TCRɑβ+ depleted cells on day of transplant (Day 0) and HPC,A infusion of CD45RA+ depleted cells on Day +1 following transplant.
  Other Names: Transplant
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System
Drug: Sirolimus — Given orally (PO) starting Day 0. The dose will be tapered off over two weeks starting on Day +42 in the absence of GVHD.
  Other Names: Rapamycin; Rapamune®

SUMMARY:
This study seeks to examine treatment therapy that will reduced regimen-related toxicity and relapse while promoting rapid immune reconstitution with limited serious graft-versus-host-disease (GVHD) and also improve disease-free survival and quality of life. The investigators propose to evaluate the safety and efficacy of selective naive T-cell depleted (by TCRɑβ and CD45RA depletion, respectively) haploidentical hematopoietic cell transplant (HCT) following reduced intensity conditioning regimen that avoids radiation in patients with hematologic malignancies that have relapsed or are refractory following prior allogeneic transplantation.

PRIMARY OBJECTIVE:

* To estimate engraftment by day +30 post-transplant in patients who receive TCRɑβ-depleted and CD45RA-depleted haploidentical donor progenitor cell transplantation following reduced intensity conditioning regimen without radiation.

SECONDARY OBJECTIVES:

* Assess the safety and feasibility of the addition of Blinatumomab in the early post-engraftment period in patients with CD19+ malignancy.
* Estimate the incidence of malignant relapse, event-free survival, and overall survival at one-year post-transplantation.
* Estimate incidence and severity of acute and chronic (GVHD).
* Estimate the rate of transplant related mortality (TRM) in the first 100 days after transplantation.

DETAILED DESCRIPTION:
Blood progenitor cells will be obtained from a partially matched adult family member (donor). After processing and filtration using the CliniMACS device, cells will be infused into participants meeting eligibility criteria.

Prior to transplant, participants will receive a conditioning treatment of rabbit ATG, cyclophosphamide, fludarabine, thiotepa, melphalan, and rituximab. Mesna will be given to help prevent side effects of cyclophosphamide. Tacrolimus will be given to help reduce the risk of GVHD. G-CSF will be given after transplant to help the donor progenitor cells make white blood cells faster so that the immune system is better able to fight infection.

Blood progenitor cells will be given in two infusions on Day 0 and Day +1. Progenitor cells then move through the blood stream to the bone marrow space where they should begin to grow. Participant blood will be monitored for 100 days to assure that the progenitor cells begin to grow. If the growth is low, additional progenitor cells may be given.

Blood tests will be monitored for up to one year to observe how well the donor cells grow and their effect on the infection-fighting system.

ELIGIBILITY:
Inclusion Criteria for Transplant Recipient:

* Age less than or equal to 21 years.
* Any of the following hematologic malignancies that has relapsed or remains refractory after prior allogeneic HCT (this includes any stage of disease - such as refractory due to induction failure, refractory in relapse, or in any CR - as long as the hematologic malignancy remained persistent or returned after a previous allogeneic HCT):

  * ALL, AML, Myeloid Sarcoma, CML, Juvenile myelomonocytic leukemia (JMML), myelodysplastic syndrome (MDS), non-Hodgkin lymphoma (NHL)
* Has a suitable single haplotype matched (≥ 3 of 6) family member donor.
* Does not have any other active malignancy other than the one for which this transplant is indicated.
* If prior CNS leukemia, it must be treated and in CNS CR
* Does not have current uncontrolled bacterial, fungal, or viral infection.
* There is no minimum time from the previous transplant, but patients must meet the following criteria:

  * Left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%.
  * Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2.
  * Forced vital capacity (FVC) ≥ 40% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing.
  * Karnofsky or Lansky (age-dependent) performance score ≥ 50 (See Appendix A).
  * Bilirubin ≤ 3 times the upper limit of normal for age.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age.
  * Not pregnant. If female with child bearing potential, must be confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
  * Not breast feeding

Inclusion Criteria for Haploidentical Donor:

* At least single haplotype matched (≥ 3 of 6) family member
* At least 18 years of age.
* HIV negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.
* Regarding donation eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients engrafted by day +30 post-transplant | 30 days post-transplant
  ANC engraftment is defined as the first of 3 consecutive tests performed on different days of an ANC ≥ 500/mm^3 with evidence of donor cell engraftment.

SECONDARY OUTCOMES:
The number of patients experiencing Blinatumomab permanent discontinuation due to toxicity | 3 months post-transplant
  If the drug is held for more than 2 weeks due to toxicity, it will be permanently discontinued.
The estimate of cumulative incidence of relapse | One year post-transplant
  The estimate of cumulative incidence of relapse will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The Kaplan-Meier estimates of overall survival (OS) and event-free survival (EFS) along with their standard errors will be calculated.
  OS is defined as time from transplantation to death or last follow-up, whichever comes first. EFS is defined as time from transplantation to events including relapse, graft failure, death due to any cause and last follow-up whichever comes first. The participants surviving at the time of analysis without events will be censored.
The cumulative incidence of acute and chronic Graft-Versus-Host Disease (GVHD) | One year post transplant
  The cumulative incidence of acute and chronic GVHD will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. GVHD will be reported separately for participants receiving tacrolimus and those receiving sirolimus.
  The severity of acute GVHD and chronic GVHD will be described.
The cumulative incidence of transplant related mortality | 100 days post transplant
  The cumulative incidence of transplant related mortality will be estimated using Kalbfleisch-Prentice method. Deaths before day 100 because of other reasons are the competing risk events.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols